CLINICAL TRIAL: NCT02725762
Title: A Double-Masked, Randomized, Sham-Controlled, Parallel Group, Single-Center Study to Assess the Safety and Efficacy of Photobiomodulation in Subjects With Dry Age-Related Macular Degeneration
Brief Title: Study of Photobiomodulation to Treat Dry Age-Related Macular Degeneration
Acronym: LIGHTSITE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LumiThera, Inc. (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSP001; 1R43EY025508-01 (NIH)
Record Dates: First submitted 2016-03-23; First posted 2016-04-01 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Age Related Macular Degeneration
Keywords: Dry AMD; Vision Loss; AMD
MeSH Terms: conditions — Macular Degeneration; Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Photobiomodulation Treatment (Experimental): Treatment with Photobiomodulation to the retina at specific wavelengths to the eye three times a week for three weeks, repeated at six months.
  Interventions: Device: LT-300 Active (PBM)
- Sham Treatment (Sham Comparator): Sham treatment to the retina at specific wavelengths to the eye three times a week for three weeks, repeated at six months.
  Interventions: Device: LT-300 Inactive (Sham)

INTERVENTIONS:
Device: LT-300 Active (PBM)
  Arms: Photobiomodulation Treatment
Device: LT-300 Inactive (Sham)
  Arms: Sham Treatment

SUMMARY:
The purpose of this research study is to determine if photobiomodulation is an effective treatment of Dry Age-Related Macular Degeneration (AMD) and vision loss associated with the disease.

DETAILED DESCRIPTION:
The LumiThera LT 300® Light Delivery System is a stationary desktop instrument used to emit energy in the visible and near infrared spectrum. The LT-300® is designed for the ophthalmologist to use in the treatment of the eye with photobiomodulation (PBM), a process by which cellular mechanisms are induced by light. PBM is being utilized in many indications, such as wound healing, soft tissue injuries, joint pain, myofascial pain, nerve injuries, muscle fatigue for temporary improvement in blood flow and reduction in inflammation. The mechanism of PBM at the cellular level has been ascribed to the activation of mitochondrial respiratory chain components resulting in stabilization of metabolic function and initiation of a signaling cascade, which promotes cellular proliferation and cytoprotection. The LT-300® will provide a preset treatment of PBM to the subject's eye and retinal tissue through the open and closed eyelid.

Approximately 30 subjects meeting the eligibility requirements of the study will be randomly assigned in a 1:1 ratio to receive standard of care treatment for Dry AMD plus PBM treatment with the LT-300 system, or standard of care treatment for Dry AMD plus Sham treatment with the LT-300 system. Subjects randomized to each group will receive two 3-week treatment sessions (9 treatments per session) and follow-up visits extending to one year. The primary objective of the study is to evaluate the safety and efficacy of PBM with respect to visual and anatomical outcomes of subjects with Dry AMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both gender
* Patients must have dry macular degeneration in the study eye
* Best corrected visual acuity between 20/40 and 20/200
* Patients must be competent to sign and have signed a consent form before study entry

Exclusion Criteria:

* Visually significant cataracts.
* Presence of a visually significant posterior capsule if prior cataract surgery has been performed.
* Any visually significant disease process in any ocular structure that would affect vision unrelated to macular degeneration.
* A patient can be enrolled if only one of their eyes meets the criteria. The other eye may be treated but not included in the study; for example advanced geographic atrophy.
* Patients with severe clinically significant disease or unstable medical disorders including cardiovascular, hepatic, renal, neurological, endocrine, gastrointestinal, CNS or life threatening disease or current malignancy at the discretion of the investigators
* Patients who are non-ambulatory or bed ridden
* Female patients who are pregnant or of childbearing potential as effects of PBM on the developing human fetus are unknown.
* Patients with a history of Epilepsy
* Patients with a history of alcohol, drug or substance abuse in the past 6 months
* Patients deemed uncooperative or non compliant with the requirements of the protocol.
* Patients who have received any investigational drug or treatment within 30 days prior to study entry.
* Patients who are not competent to understand and sign consent form.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Visual Acuity changes from baseline to month 12. | Through study completion, an average of one year.
  Visual acuity will be measured using ETDRS VA letter scoring to test the difference between the sham and treatment subjects in mean change from Baseline to Month 12

SECONDARY OUTCOMES:
Contrast Sensitivity | Through study completion, an average of one year.
  Contrast Sensitivity will be measured using the FACT Contrast Sensitivity Chart to test the difference between the sham and treatment subjects in mean change from Baseline to Month 12
Optical Coherence Tomography (OCT) | Through study completion, an average of one year.
  OCT will be measured using the Spectralis SD-OCT to compare changes in dry AMD pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Markowitz, MD, Principal Investigator — Private Practice; Robert G Devenyi, MD, Principal Investigator — Ophthalmologist in Chief and Director of Retinal Services, The Donald K. Johnson Eye Center, University Health Network; Professor of Ophthalmology, The University of Toronto; Vitreoretinal Surgery Lead, The Kensington Eye Institute
Locations (1):
- 1929 Bayview Avenue, Unit 117, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: LIGHTSITE I Results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7392581/